CLINICAL TRIAL: NCT02423226
Title: Phase II Study of Computed Tomography-guided Brachytherapy Plus Chemotherapy for Locally Recurrent Rectum Cancer
Brief Title: Computed Tomography-guided Brachytherapy Plus Chemotherapy for Locally Recurrent Rectum Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Principal Investigator, Liangrong Shi, Director of Science and Education Division, The First People's Hospital of Changzhou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZ-I125-001
Record Dates: First submitted 2015-04-16; First posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Rectum Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Brachytherapy; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CT alone (Active Comparator): Treated with systemic chemotherapy alone (FOLFIRI).
  Interventions: Drug: Systemic chemotherapy (FOLFIRI)
- CT+BT (Experimental): Treated with systemic chemotherapy (FOLFIRI) plus computed tomography guided radioactive seeds implant.
  Interventions: Procedure: Computed tomography guided radioactive seeds implant; Drug: Systemic chemotherapy (FOLFIRI)

INTERVENTIONS:
Procedure: Computed tomography guided radioactive seeds implant — Computed tomography guided radioactive seeds implant were performed one week before chemotherapy.
  Other Names: Brachytherapy
  Arms: CT+BT
Drug: Systemic chemotherapy (FOLFIRI) — irinotecan 180mg/m2 d1,leucovorin 400mg/m2 d1, 5-fluorouracil 400mg/m2 iv, 2.4g/m2 civ 46h, repeated every 2 weeks
  Other Names: FOLFIRI

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of CT guided 125I seeds implant plus systemic chemotherapy for locally recurrent rectum cancer.

DETAILED DESCRIPTION:
The primary aim of this study is to determined the safety and efficacy of CT guided 125I seeds implant plus systemic chemotherapy for locally recurrent rectum cancer.The patients with recurrence in pelvic or on pelvic wall after rectal resection were treated with 125I seeds implant plus chemotherapy or chemotherapy alone. The side-effect, tumor response and survival data were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Limited locoregional recurrence including solitary recurrence at primary tumor bed, solitary intraabdominal peritoneal recurrence, and single regional lymph node recurrence (no more than 3 lymph nodes) based on diagnosis by CT, and confirmed by percutaneous puncture biopsy
* Second-line treatment for advanced colorectal cancer,irinotecan was not previously used.
* Age range 18-70 years old
* ECOG performance status 0-1
* Life expectancy of more than 3 months
* Adequate organ function

Exclusion Criteria:

Previous serious cardiac disease

* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Pregnant or lactating women
* Chronic inflammatory bowel disease or intestinal obstruction
* Serious uncontrolled diseases and intercurrent infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-10; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Progression free survival | One year
  Progression free survival which is calculated from the start of treatment to disease progression or death

SECONDARY OUTCOMES:
Treatment related adverse events | Eight weeks
  Including chemotherapy related side-effect and brachytherapy related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Changping Wu, M.D., Study Director — The First People's Hospital of Changzhou